CLINICAL TRIAL: NCT07326098
Title: Efficacy of Ultrasound-Guided Genicular Nerve Block in Patients With Gonarthrosis: A Randomized, Placebo-Controlled, Double-Blind Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-5.1/20
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gonarthrosis; Primary
Keywords: gait parameters; genicular nerve block; Gonarthrosis; GNB; pedogait
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — triamcinolone hexacetonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The study is conducted as a randomized, double-blind, placebo-controlled trial. Both participants and care providers administering the injections are blinded to group assignments. Syringes are prepared and covered by an independent researcher to ensure identical appearance across groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Ultrasound-guided genicular nerve block will be performed using a combination of 4 mL Priloc 2% (lidocaine) and 1 mL Artropan 20 mg (triamcinolone hexacetonide).
  The syringe's outer part will be covered by an independent researcher to conceal the contents.
  All participants will also perform a home exercise program: quadriceps strengthening and knee isometric exercises.
  Interventions: Procedure: genicular nerve block
- Placebo group (Placebo Comparator): A placebo injection with 5 mL saline solution will be administered under the same sterile and ultrasound-guided conditions.
  The syringe's outer part will be covered by an independent researcher to conceal the contents.
  All participants will also perform a home exercise program: quadriceps strengthening and knee isometric exercises.
  Interventions: Procedure: Placebo injection (normal saline)

INTERVENTIONS:
Procedure: genicular nerve block — Genicular nerve block performed with pharmacological agents under ultrasound guidance is minimally invasive compared to other block techniques. It can be carried out in an outpatient setting with attention to sterility, does not involve radiation, does not require procedural surgical preparations, and is less costly both for the patient and the healthcare system. Furthermore, it has fewer side effects, with many studies reporting no side effects at all.
  Other Names: Ultrasound-guided genicular nerve block including the combination of lidocaine and triamcinolone hexacetonide
  Arms: İntervention group
Procedure: Placebo injection (normal saline) — A placebo injection with 5 mL saline solution will be administered under the same sterile and ultrasound-guided conditions as the active group.
  The syringe will be covered by an independent researcher to conceal the contents, ensuring identical appearance across groups.
  All participants will also perform a home exercise program: quadriceps strengthening and knee isometric exercises.
  Arms: Placebo group

SUMMARY:
This study planned to enroll a minimum of 30 patients aged 50 years and older, with a diagnosis of gonarthrosis classified as stage 2 or higher according to the Kellgren-Lawrence grading system, and who report complaints of knee pain and walking difficulties. Patients will be randomized into two groups, and they will be blinded to the group to which they are assigned.

In the first group, ultrasound-guided genicular nerve block will be performed using a combination of lidocaine and triamcinolone hexacetonide injection (4 mL Priloc 2% + 1 mL Artropan 20 mg). In the second group, a placebo injection (5 mL saline solution) will be administered. Both groups will be instructed to follow an appropriate exercise program after the treatment.

Patients will undergo a detailed physical examination, 6-minute walk test, VAS pain score, WOMAC questionnaire, and 3D kinematic gait analysis with pressure parameters evaluated by a blinded researcher. Evaluations will take place before treatment, 1 hour after treatment, and 1 month post-treatment.

The collected data will be analyzed for differences between the two groups and changes over time. The potential positive effects of the treatment will be measured and compared with the placebo group to assess the therapeutic efficacy.

DETAILED DESCRIPTION:
In addition to the fact that genicular nerve block is highlighted in the literature as a potential alternative to surgery, it is also crucial to consider the reality that the pain symptoms in these patients have a more significant negative impact on walking than initially expected, potentially creating a comorbidity of its own. Given this, this study aims to contribute to the medical literature by observing the improvement in walking parameters secondary to the reduction of pain symptoms in patients with gonarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain persisting for 3 months or longer
* Diagnosis of gonarthrosis with Grade 2 or higher tibiofemoral osteoarthritis detected on plain radiographs
* Patients aged 50 years and older
* Continued pain despite conservative treatment (exercise, simple analgesics such as paracetamol, or nonsteroidal anti-inflammatory drugs)

Exclusion Criteria:

* Clinical diagnoses that could cause knee pain other than gonarthrosis (rheumatologic diseases, secondary osteoarthritis, fractures, etc.)
* Signs of inflammation/exacerbation
* Infection at the injection site or skin lesions
* Diagnosis of malignancy
* Gait impairment (the patient must be able to ambulate independently)
* Known allergy to study medications
* Previous knee surgery
* Uncontrolled comorbid conditions such as diabetes mellitus or hypertension, which contraindicate corticosteroid use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect on gait kinematics | 4 weeks
  Change in gait and pressure parameters measured with the DIERS Formetric 4D analysis system.
1. 6 minute walk test | 4 weeks
  It is a test used to assess the level of functional exercise or functional capacity. The patient is asked to walk, but not run, in a 25 m long corridor at the highest possible speed without stopping. At the end of 6 minutes, the number of metres walked by the patient is recorded. The 6 min walk test is an evaluation criterion used in routine and clinical research to assess functional capacity in many diseases such as heart failure, general arthrosis, multiple sclerosis.

SECONDARY OUTCOMES:
(VAS) for pain and fatigue | 4 weeks
  Severity of pain that the participants have had in the past week was evaluated by using visual analogue scale (VAS) on a 10-cm horizontal line where 0-cm represented "no pain" and 10 cm the "worst imaginable pain" Severity of fatigue experienced by the participants in the past week was assessed by using VAS on a 10-cm horizontal line where 0-cm represented "not tired at all" and 10-cm "extremely tired"
WOMAC | 4 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a valid and reliable questionnaire frequently used in clinical and research settings for patients with knee osteoarthritis. It consists of 24 questions and includes three subcategories: pain, stiffness, and physical function. The patient fills out the questionnaire themselves. The pain subcategory is assessed with five questions, stiffness with two questions, and physical function with 17 questions. Each question is scored according to a Likert scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. The subcategories are evaluated independently. Higher scores on the questionnaire indicate a greater degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Cinar, Assistant Professor, Principal Investigator — EGE UNİVERCİTY
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University Faculty of Medicine, Izmir, Bornova
  - Ege University Faculty of Medicine, Izmir

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lebleu J, Fonkoue L, Bandolo E, Fossoh H, Mahaudens P, Cornu O, Detrembleur C. Lower limb kinematics improvement after genicular nerve blockade in patients with knee osteoarthritis: a milestone study using inertial sensors. BMC Musculoskelet Disord. 2020 Dec 7;21(1):822. doi: 10.1186/s12891-020-03836-8. PMID 33287783